CLINICAL TRIAL: NCT04202536
Title: A Randomized, Open-Label, Parallel, Multi-Center, Non-inferiority, Phase IV Clinical Trial to Evaluate the Efficacy and Safety of Switching to Besifovir Dipivoxil Maleate From Tenofovir Disoproxil Fumarate (TDF) in Chronic Hepatitis B Patients Who Pretreated With TDF
Brief Title: Switching From Tenofovir Disoproxil Fumarate to Besifovir Dipivoxil Maleate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID-BVCL-403
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B; Besifovir Dipivoxil Maleate; Tenofovir Disoproxil Fumarate
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TDF switch to Besifovir Dipivoxil Maleate (Experimental): Tenofovir Disoproxil Fumarate(TDF) 300mg daily switch to Besifovir Dipivoxil Maleate 183mg daily
  Interventions: Drug: Besifovir Dipivoxil Maleate
- Maintaining on TDF (Active Comparator): Maintaining on Tenofovir Disoproxil Fumarate(TDF) 300mg daily
  Interventions: Drug: Tenofovir disoproxil fumarate(TDF)

INTERVENTIONS:
Drug: Besifovir Dipivoxil Maleate — Besifovir 150 mg q.d. + L-carnitine (L-Carn Tab. 330 mg) 660 mg q.d. Other Name: Besifovir®
  Arms: TDF switch to Besifovir Dipivoxil Maleate
Drug: Tenofovir disoproxil fumarate(TDF) — 300 mg tablet administered orally once daily Other Name: VIREAD®
  Arms: Maintaining on TDF

SUMMARY:
A research study to observe the safety, efficacy and tolerability of switching from Tenofovir Disoproxil Fumarate to Besifovir dipivoxil maleate in patients with chronic hepatitis B

ELIGIBILITY:
Inclusion Criteria:

1. 20 years of age and older, Male or female patients
2. Patients who show positive HBsAg or has a history of chronic hepatitis B for the last six months or more before screening
3. Patients who have been on tenofovir disoproxil fumarate (TDF) monotherapy for more than 48 weeks and are taking TDF at the time of clinical screening
4. At screening, had HBV DNA < 20 IU/mL
5. Patients who were explained about the purpose, methods and effects of the clinical trial and then, signed a written consent form

Exclusion Criteria:

1. Patients who have received interferon (including Pegylation formulation) to treat chronic hepatitis for more than 12 months.
2. Patients who have taken Besifovir
3. Patients who have experienced hepatitis B virus resistance to antiviral drugs
4. Patient diagnosed with a malignant tumor within 5 years before screening or relapsed patient
5. Patient has history of organ transplantation
6. Patients who had received the following drugs for the last two months before screening (however, short-term use (less than consecutive 14 days) of these drugs and low-dose aspirin (100 mg, maximally, 300 mg/day) are allowed.)

   * Nephrotoxic drugs (e.g. Aminoglycosides, Amphotericin B, NSAIDs)
   * Hepatotoxic drugs (e.g. Erythromycin, Ketoconazole, Rifampin, Fluconazole, Dapsone)
   * Anticoagulant (e.g. Warfarin)
7. Patients who are suspected by an investigator to have the level of immunity decreased among patients who had been administered with immunosuppressants within 12 months before screening
8. Patients who had been administered with long-term general corticosteroids (more than consecutive 14 days) at a high dose (more than prednisolone 20 mg daily*) within three months before screening (In case of local corticosteroids, an investigator decides it.)

   * It is equal to cortisone 125 mg, hydrocortisone 100 mg, prednisone 20 mg, methylprednisolone 16 mg, triamcinolone 16 mg, dexamethasone 3 mg, betamethasone 2.4 mg
9. Patients who have a past medical history of clinical alcohol or drug abuse within a year before screening or now are abusers
10. Patients with hepatitis C virus, hepatitis D virus or human immunodeficiency virus
11. Patients who have other hepatic diseases (hematochromatosis, Wilson's disease, alcoholic liver diseases, nonalcoholic steatohepatitis, α1-antitrypsin deficiency) except hepatitis B
12. Patient concerned about the decline in daily activity or not able to understand the objectives and methods due to the psychiatric problems
13. Patients who showed Glomerular Filtration Rate (GFR) less than 50 mL/min by calculating Modification of Diet in Renal Disease (MDRD: 1.86 x phosphocreatine -1.154 x age -0.203 (x 0.742 for women)) during screening
14. Patients who showed alpha-fetoprotein(AFP) more than 50 ng/mL during screening and are estimated to have hepatocellular carcinoma (HCC) through liver/abdomen CT scans
15. At least one of the following laboratory values during screening

    * Hemoglobin < 9.0 g/dL
    * Absolute neutrophil count (ANC) < 1.0 x 10^9 /L (1000 /mm^3)
    * Platelet count < 75 x 10^9 /L (100 x 10^3 /mm3)
    * Serum creatinine > 1.5 mg/dL
    * Serum amylase > 2 x upper limit normal (ULN) and Lipase > 2 x ULN
    * Total Bilirubin > 2 x ULN
    * Serum albumin < 28 g/L (2.8 g/dL)
16. Pregnant women, lactating women, or patients who planned pregnancy during a trial period
17. Patients who participate in other clinical trials or is supposed to do so during the study period
18. Patients who have hypersensitivity to the clinical trial drug in this clinical trial
19. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
20. Patients who are considered to be unacceptable in this study under the opinion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The rate of subjects who maintained hepatitis B virus (HBV) DNA less than 20 IU/mL at the 48th week | at the 48th week

SECONDARY OUTCOMES:
The rate of subjects who maintained HBV DNA less than 20 IU/mL at the 24th week | at the 24th week

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Medical Center, Ansan, Kyounggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No